CLINICAL TRIAL: NCT03530657
Title: the Department of Medical Ultrasound, Third Affiliated Hospital of Sun Yat-Sen University
Brief Title: Assessment of Liver Fibrosis and Prognosis in Chinese Patients With CHB Infection Using STE/STQ Elastography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Rongqin Zheng, the Department of Medical Ultrasound, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: STE/STQ 2018
Record Dates: First submitted 2018-04-20; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Liver biopsy specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This national multicenter prospective study is aimed to study the diagnositic performance of STE/STQ elastography in liver fibrosis and prognosis in patients with chronic hepatitis B infection.

DETAILED DESCRIPTION:
Ultrasound liver elasticity measurement and imaging has not only been proposed as an alternative to evaluate the severity of chronic liver fibrosis, but also as a mean to stratify patients with advanced fibrosis according to risks of occurrence of clinical complications of end-stage liver diseases.

Sound touch elastography (STE）and sound touch quantify (STQ) developed by Mindray Resona 7 imaging system provide both two-dimensional and point shear-wave elastography of tissue elasticity with stronger penetration and easy operation.

This analysis will study the diagnositic performance of STE/STQ elastography for lver fibrosis and the prognostic value of STE/STQ elastography for the prediction of clinical complications of chronic liver diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a liver ultrasound exam due to confirmed Hepatitis B infection ,
* Patients having reached the age of majority in China,
* Patients with a liver biopsy for histological evaluation of liver fibrosis, performed within 3 months after the STE/STQ measurement date, and having the recommended quality criterion:

minimal length of biopsy samples of 15 mm, stored in paraffin minimal number of portal tracts of 6 per biopsy samples

* Patients of Chinese ethnic origin.

Exclusion Criteria:

Any of the conditions below will exclude patients from the study:

* Any patient presenting with combined etiologies of chronic liver diseases:，including Non hepatitis B viral infection（Hepatitis A, C, D, E）, alcoholic chronic liver disease, hemochromatosis, autoimmune hepatitis，etc
* Any patient presenting with a co-infection of HIV
* Any patient presenting with combined liver tumor
* Any patient ever received liver transplantation
* Pregnant women
* Acute hepatitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are recruited from primary care clinic
Sampling Method: Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2018-06-04 (Estimated); Primary Completion 2020-06-04 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Degree of Liver Fibrosis | 1-2 years
  All liver biopsies will be taken for evaluating the degree of liver fibrosis according to the METAVIRE classification. The degree of fibrosis is classified in a 0-4 scale as follows: F0: no fibrosis, F1: portal fibrosis alone, F2: portal fibrosis with rare septa, F3: portal fibrosis with many septa, and F4: cirrhosis.

SECONDARY OUTCOMES:
Complication rates depending on liver STE/STQ measurement values at baseline | 2 years
  Clinical complications in our study protocol are: ascites, hepatic encephalopathy, esophageal varices, fundal varices, variceal bleeding, liver failure, HCC and death. The complication rates are regarded as occurrence of clinical complications in patients with chronic hepatitis B.